CLINICAL TRIAL: NCT00967044
Title: Phase I/II of Panobinostat (LBH589) Plus Everolimus (RAD001) in Patients With Relapsed and Refractory Lymphoma
Brief Title: Panobinostat (LBH589) Plus Everolimus (RAD001) in Patients With Relapsed and Refractory Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0805; NCI-2011-03023 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Lymphoma
Keywords: Relapsed or Refractory Lymphoma; Hodgkin's lymphoma; Non Hodgkin's Lymphoma; NHL; LBH589; Panobinostat; RAD001; Everolimus
MeSH Terms: conditions — Lymphoma; Recurrence; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Panobinostat; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panobinostat + Everolimus (Experimental): Panobinostat (LBH589) Plus Everolimus (RAD001)
  Interventions: Drug: Panobinostat; Drug: Everolimus

INTERVENTIONS:
Drug: Panobinostat — Starting dose of 10 mg by mouth per day, self-administered (by patients), three times per week
  Other Names: LBH589
Drug: Everolimus — Starting dose of 5 mg every day by mouth with 1 cup (8 ounces) of water, in morning after eating a low-fat meal.
  Other Names: Afinitor; RAD001

SUMMARY:
Objectives:

Primary:

* Determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of the novel combination of everolimus + Panobinostat (LBH589) in a phase-I study in patients with relapsed lymphoma (Hodgkin and non-Hodgkin).
* Determine the safety and efficacy of this novel combination in a phase-II study in patients with relapsed Hodgkin and non-Hodgkin lymphoma

Secondary:

* Determine the in vivo effect of therapy on selected serum cytokines/chemokines (TGF-beta, thymus and activation-regulated chemokine (TARC), IL-6, IL-10, VEGF).
* Examine pre-treatment level of selected molecular targets (HDACs 1-11, STAT6, pSTAT6, STAT3, pSTAT3, Myc, Akt, Pichia anomala killer toxin (pAkt), S6, pS6, p21, cyclin D1) in primary lymphoma cells and the surrounding reactive inflammatory cells obtained by core needle biopsies from patients with relapsed lymphoma.
* Examine the correlation between molecular and biologic markers and clinical response and/or treatment-related toxicity.

DETAILED DESCRIPTION:
Phase I:

The Study Drugs:

Both panobinostat and everolimus are designed to block cancer cells from multiplying. Everolimus may also stop the growth of new blood vessels that help tumor growth. As a result, the cancer cells may grow more slowly or die.

Study Groups:

If you are found to be eligible to take part in this phase of the study, you will be assigned to a study group based on when you joined this study. Up to 5 groups of 3-6 participants will be enrolled in this phase of the study.

If you are enrolled in this phase of the study, the dose of study drugs you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of the study drugs. Each new group may receive a higher dose of study drugs than the group before it, if no intolerable side effects were seen. This will continue for up to 5 combinations of the study drugs, until the highest tolerable dose of study drugs in combination is found.

Up to 2 dose levels of everolimus and up to 4 dose levels of panobinostat will be tested in this phase of the study. This is up to 5 different dose combinations of everolimus and panobinostat. (The dose of both drugs does not get raised in every dose level, but sometimes only 1 drug's dose gets raised.)

Study Drug Administration:

Panobinostat:

You will take panobinostat by mouth 3 times a week during each cycle. Cycles in this study are 28 days long.

You should take panobinostat with 1 cup (8 ounces) of water at about the same time each day that you take it.

If you miss a dose of panobinostat, take it as soon as you remember it on the same day. However, if more than 12 hours have passed since you were supposed to take the dose, you should skip that day's dose. In that case, wait to take panobinostat until the next scheduled treatment day.

Everolimus:

You will take everolimus every day, at about the same time in the morning. You will take it by mouth with 1 cup (8 ounces) of water. You should take everolimus either with no food or drink except water ("fasting") or with no more than a light, fat-free meal.

Examples of light, fat-free meals include cereal with fat-free milk, a fat-free muffin, toast, a bagel with fat-free spread, or fruit salad.

The reason to avoid high-fat breakfasts while you are taking everolimus is to help the drug get absorbed better by your body.

If you experience intolerable side effects, you must call your doctor right away. The doctor may then lower the dose of study drug or take you off study.

You should not consume grapefruit products or Seville (sour) oranges while you are on study, because they may interact with everolimus.

Study Visits:

Within 7 days before the first dose of study drug:

* You will be asked about any drugs you may be taking.
* Blood (about 2 1/2 teaspoons) and urine will be collected for routine tests.
* Women who are able to become pregnant will have a blood (about 1 tablespoon) pregnancy test.

On Day 1 of Cycle 1:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects that may have occurred.
* Your performance status will be recorded.
* Blood (about 2 1/2 teaspoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) will be drawn for biomarker research.
* If your doctor thinks it is needed, urine will be collected for routine tests.
* Women who are able to become pregnant will have a blood (about 1 tablespoon) pregnancy test.

On Days 1 and 5 of Cycle 1, you will have an ECG.

On Weeks 2, 3, and 4 of Cycle 1, blood (about 2 1/2 teaspoons) will be drawn for routine tests.

On Week 2 of Cycle 1, blood (about 1 teaspoon) will be drawn for biomarker research.

On Day 1 of Cycle 2 and every cycle after that:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects that may have occurred.
* Your performance status will be recorded.
* You will have an ECG (or more than 1 ECG if the doctor thinks it is needed).
* Blood (about 2 1/2 teaspoons) will be drawn for routine tests.
* Women who are able to become pregnant will have a blood (about 1 tablespoon) pregnancy test.

Every 8 weeks:

* You will have a PET scan to check the status of the disease.
* You will have a CT scan of your head and neck, chest, abdomen, and pelvis to check the status of the disease.

Length of Study:

If you show benefit from taking the study drugs, you may receive up to 6 cycles. You will be taken off study if you have intolerable side effects or the disease gets worse.

End-of-Treatment Visit:

After you stop taking the study drugs, you will return to the clinic for an end-of-treatment visit:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will have an ECG.
* You will be asked about any drugs you may be taking.
* Blood (about 3 1/2 teaspoons) will be collected for routine tests.
* You will have a PET scan to check the status of the disease.
* You will have a computed tomography (CT) scan of your head and neck, chest, abdomen, and pelvis to check the status of the disease.
* If your doctor thinks it is needed, urine will be collected for routine tests.
* If the doctor thinks the disease has responded completely, you will have a bone marrow biopsy and aspiration to confirm the complete response. To collect a bone marrow biopsy/aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.
* Women who are able to become pregnant will have a blood (about 1 tablespoon) pregnancy test.

This is an investigational study. Panobinostat is not FDA approved or commercially available. At this time the drug is being used in research only. Everolimus is FDA approved and commercially available for the treatment of renal cell carcinoma. Using everolimus in combination with panobinostat in patients with lymphoma is investigational.

Up to 18 patients will take part in this phase of this study. All will be enrolled at MD Anderson.

Phase II:

The Study Drugs:

Both panobinostat and everolimus are designed to block cancer cells from multiplying. Everolimus may also stop the growth of new blood vessels that help tumor growth. As a result, the cancer cells may grow more slowly or die.

Study Drug Administration:

Panobinostat:

You will take panobinostat by mouth 3 times a week during each cycle. Cycles in this study are 28 days long.

You should take panobinostat with 1 cup (8 ounces) of water at about the same time each day that you take it.

If you miss a dose of panobinostat, take it as soon as you remember it on the same day. However, if more than 12 hours have passed since you were supposed to take the dose, you should skip that day's dose. In that case, wait to take panobinostat until the next scheduled treatment day.

Everolimus:

You will take everolimus every day, at about the same time in the morning. You will take it by mouth with 1 cup (8 ounces) of water. You should take everolimus either with no food or drink except water ("fasting") or with no more than a light, fat-free meal.

Examples of light, fat-free meals include cereal with fat-free milk, a fat-free muffin, toast, a bagel with fat-free spread, or fruit salad.

The reason to avoid high-fat breakfasts while you are taking everolimus is to help the drug get absorbed better by your body.

If you experience intolerable side effects, you must call your doctor right away. The doctor may then lower the dose of study drug or take you off study.

You should not consume grapefruit products or Seville (sour) oranges while you are on study, because they may interact with everolimus.

Study Visits:

Within 7 days before the first dose of study drug:

* You will be asked about any drugs you may be taking.
* Blood (about 2 1/2 teaspoons) and urine will be collected for routine tests.
* Women who are able to become pregnant will have a blood (about 1 tablespoon) pregnancy test.

On Day 1 of Cycle 1:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects that may have occurred.
* Your performance status will be recorded.
* Blood (about 2 1/2 teaspoons) will be drawn for routine tests.
* Blood (about 4 tablespoons) will be drawn for biomarker research (if blood was not drawn for biomarker research at screening).
* If your doctor thinks it is needed, urine will be collected for routine tests.
* Women who are able to become pregnant will have a blood (about 1 tablespoon) pregnancy test.

On Days 1 and 5 of Cycle 1, you will have an ECG.

On Weeks 2, 3, and 4 of Cycle 1, blood (about 2 1/2 teaspoons) will be drawn for routine tests.

On Weeks 2 and 3 of Cycle 1, blood (about 4 tablespoons) will be drawn for biomarker research.

On Day 1 of Cycle 2 and every cycle after that:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will be asked about any drugs you may be taking and any side effects that may have occurred.
* Your performance status will be recorded.
* You will have an ECG (or more than 1 ECG if the doctor thinks it is needed).
* Blood (about 2 1/2 teaspoons) will be drawn for routine tests.
* Women who are able to become pregnant will have a blood (about 1 tablespoon) pregnancy test.

Every 8 weeks:

* You will have a PET scan to check the status of the disease.
* You will have a CT scan of your head and neck, chest, abdomen, and pelvis to check the status of the disease.

Length of Study:

You may continue receiving the study drugs for as long as you are benefitting. You will be taken off study if you have intolerable side effects or the disease gets worse.

End-of-Treatment Visit:

After you stop taking the study drugs, you will return to the clinic for an end-of-treatment visit:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will have an ECG.
* You will be asked about any drugs you may be taking.
* Blood (about 3 1/2 teaspoons) will be collected for routine tests.
* You will have a PET scan to check the status of the disease.
* You will have a computed tomography (CT) scan of your head and neck, chest, abdomen, and pelvis to check the status of the disease.
* If your doctor thinks it is needed, urine will be collected for routine tests.
* If the doctor thinks the disease has responded completely, you will have a bone marrow biopsy and aspiration to confirm the complete response. To collect a bone marrow biopsy/aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.
* Women who are able to become pregnant will have a blood (about 1 tablespoon) pregnancy test.

This is an investigational study. Panobinostat is not FDA approved or commercially available. At this time the drug is being used in research only. Everolimus is FDA approved and commercially available for the treatment of renal cell carcinoma. Using everolimus in combination with panobinostat in patients with lymphoma is investigational.

Up to 42 patients will take part in this phase of this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Hodgkin or non Hodgkin's lymphoma
2. Relapsed or refractory after standard treatments and with no curative option with conventional therapy
3. No evidence of cerebral or meningeal involvement by lymphoma
4. Age >= 18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
6. Life expectancy of at least 3 months
7. Signed informed consent form prior to enrollment
8. Patients must meet the following laboratory criteria: Aspartate aminotransferase (AST)/serum glutamate oxaloacetate transaminase (SGOT) and ALT/serum glutamate pyruvate transaminase (SGPT) </= 2.5 * upper limit of normal (ULN) ) or </= 5.0 x ULN if the transaminase elevation is due to lymphoma involvement, Serum bilirubin </= 1.5 * ULN, Serum creatinine </=1.5 * ULN free T4 within normal limits (WNL) (patients may be on thyroid hormone replacement)
9. Patients must have at least one measurable site of disease
10. Adequate bone marrow function as shown by: Absolute neutrophil count (ANC) >/= 1.0 x 109/L, Platelets >/=100 x 109/L
11. Fasting serum cholesterol </=300 mg/dL OR </=7.75 mmol/L AND fasting triglycerides </= 2.5 * ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication 24 hours before starting therapy.
12. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study drug

Exclusion Criteria:

1. Burkitt's lymphoma, Lymphoblastic lymphoma, Chronic lymphocytic leukemia (Small lymphocytic lymphoma may be included)
2. Chemotherapy or radiation therapy or other investigational agents within 4 weeks prior to entering the study
3. Previous radioimmunotherapy within 12 weeks
4. Prior therapy with HDAC or [1] mammalian target of rapamycin (mTOR) inhibitors i.e. temsirolimus, vorinostat (the list is not inclusive of investigational agents in these classes of drugs)
5. Patient with known HIV infection
6. Known active viral hepatitis
7. Any serious active disease or co-morbid condition, which in the opinion of the principle investigator, will interfere with the safety or with compliance with the study
8. Impaired cardiac function including any one of the following: • Screening ECG with a corrected QT interval (QTc) > 450 msec confirmed by the investigator prior to enrollment to the study • Patients with congenital long QT syndrome • History of sustained ventricular tachycardia • Any history of ventricular fibrillation or torsades de pointes • Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate >= 50 beats per minute are eligible.
9. Impaired cardiac function including any one of the following continued: • Patients with a myocardial infarction or unstable angina within 6 months from registration on study • Congestive heart failure (NY Heart Association class III or IV) • Right bundle branch block and left anterior hemiblock (bifascicular block) • Uncontrolled hypertension
10. Concomitant use of drugs with a risk of causing torsades de pointes
11. Patients with unresolved diarrhea Common Toxicity Criteria for Adverse Effects (CTCAE) grade 1
12. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral PANOBINOSTAT or everolimus.
13. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception.
14. Male patients whose sexual partners are WOCBP not using effective birth control
15. Patients with a history of another primary malignancy within 5 years other than curatively treated CIS of the cervix, basal or squamous cell carcinoma of the skin, or early stage prostate carcinoma.
16. Patients with known positivity for human immunodeficiency virus (HIV) ) or hepatitis C; baseline testing for HIV and hepatitis C is not required
17. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
18. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent, except corticosteroids with a daily dosage equivalent to prednisone <= 20 mg. Topical or inhaled corticosteroids are allowed.
19. Patients should not receive immunization with attenuated live vaccines within one week of study registration or during study period
20. Chronic obstructive pulmonary disease (COPD) or asthma requiring therapy
21. Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
22. Active (acute or chronic) uncontrolled severe infection, requiring oral or intravenous antibiotics.
23. Patients receiving treatment on another clinical research trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Oki, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 25, 2009 to February 17, 2012. All recruitment was done at University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 31 participants recruited, one participant was excluded from the study as a screen failure.
Period: Overall Study
Arm/Group | Panobinostat + Everolimus
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 30 patients were evaluated in intention to treat based response analysis.
Groups:
- Panobinostat + Everolimus: Panobinostat (LBH589) Plus Everolimus (RAD001)
  Panobinostat: Starting dose of 10 mg by mouth per day, self-administered (by participants), three times per week.
  Everolimus: Starting dose of 5 mg every day by mouth with 1 cup (8 ounces) of water, in morning after eating a low-fat meal.
Arm/Group | Panobinostat + Everolimus
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 52 [20 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 30
Participation by Cohort [Number; unit: participants] — Participant by Cohort (1 to 4) according to Panobinostat dose (mg/orally taken three times weekly) and Everolimus dose (mg/orally taken daily).
  participants
    Panobinostat 10 mg/Everolimus 5 mg | 3
    Panobinostat 20 mg/Everolimus 5 mg | 3
    Panobinostat 20 mg/Everolimus 10 mg | 22
    Panobinostat 30 mg/Everolimus 10 mg | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Everolimus With Panobinostat
Description: MTD of the novel combination of Everolimus + Panobinostat (LBH589) in a phase-I study in participants with relapsed lymphoma (Hodgkin and non-Hodgkin) where MTD is defined as the highest dose at which no more than 1 in 6 of the participants in the cohort experiences one or more dose limiting toxicities (DLTs) in the first 28 day treatment cycle. Thirty patients were enrolled onto four dose levels: Everolimus (mg, orally) 5, 5, 10, 10 daily or Panobinostat (mg, orally) 10, 20, 20, 30 three times per week. The MTD was established without the use of colony stimulating factor in cycle 1.
Time Frame: 28 day treatment cycle
Measure: Number; unit: mg, orally
Arm/Group | Panobinostat + Everolimus
Number analyzed (Participants) | 30
mg, orally
  Everolimus (daily) | 10
  Panobinostat (three times weekly) | 20

ADVERSE EVENTS:
Time Frame: Adverse event reporting with each 28 day treatment cycle. Overall study participation from December 2009 to April 2012.
Arm/Group | Panobinostat + Everolimus
Serious Adverse Events (participants affected / at risk) | 19/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat + Everolimus (N=30)
Fatigue (General disorders) | 2 (2) — Grade 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Grade 3
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 3
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) — Grade 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) — Grade 4
Febrile neutropenia (Infections and infestations) | 2 (2) — Grade 3
Other Infection (Infections and infestations) | 3 (3) — Two Grade 3, One Grade 4
Anemia (Blood and lymphatic system disorders) | 6 (6) — Four Grade 3, Two Grade 4
Neutropenia (Blood and lymphatic system disorders) | 14 (14) — Nine Grade 3, Five Grade 4
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (19) — Two Grade 3, Seventeen Grade 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat + Everolimus (N=30)
Anorexia (General disorders) | 17 (17)
Weight loss (General disorders) | 10 (10)
Fatigue (General disorders) | 25 (25)
Dizziness (General disorders) | 6 (6)
Edema (General disorders) | 8 (8)
Nausea (General disorders) | 10 (10)
Vomit (General disorders) | 3 (3)
Pain (General disorders) | 12 (12)
Rigors (General disorders) | 5 (5)
Hypotension (Cardiac disorders) | 6 (6)
QTc prolongation (Cardiac disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Elevated ALKP (Gastrointestinal disorders) | 5 (5) — serum alkaline phosphatase (ALKP)
Elevated AST (Gastrointestinal disorders) | 8 (8) — serum aspartate aminotransferase (AST)
Diarrhea (Gastrointestinal disorders) | 14 (14)
Mucositis (Gastrointestinal disorders) | 18 (18)
Hyperglycemia (Metabolism and nutrition disorders) | 19 (19)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesiemia (Metabolism and nutrition disorders) | 5 (5)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 10 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Dysphasia (Nervous system disorders) | 3 (3)
Sensory neuropathy (Nervous system disorders) | 8 (8)
Taste change (Nervous system disorders) | 7 (7)
Elevated creatinine (Renal and urinary disorders) | 6 (6)
Acne (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 10 (10)
Rhinitis (Ear and labyrinth disorders) | 7 (7)
Non-neutropenic fever (Infections and infestations) | 10 (10)
Other infection (Infections and infestations) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 16 (16)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hemorrhage (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Initially intended to proceed to phase II at MTD, treatment interruptions were frequently required in participants treated at MTD for Grade 3/4 Thrombocytopenia so study amended to obtain more detailed safety data at MTD in expanded phase I study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No